CLINICAL TRIAL: NCT03251755
Title: The Effectiveness of Dao-in (Chinese Yoga) on Insomnia in Type 2 Diabetes Mellitus
Brief Title: Exercise Using Chinese Yoga Improving Insomnia
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Deputy head nurse, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE17071B
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Exercise Promotion
Keywords: type 2 diabetes mellitus; insomnia; Dao-in
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Open-labelled, randomized, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise promotion using Dao-in (Chinese Yoga)
  Interventions: Behavioral: Yoga
- Control (No Intervention): Usually clinical practice

INTERVENTIONS:
Behavioral: Yoga — Exercise promotion using Chinese Yoga
  Arms: Exercise

SUMMARY:
According to the data from WHO, currently there are 350 million people with diabetes mellitus in the world, and the amount of which is still increasing. Among all types of diabetes mellitus, people with type 2 diabetes mellitus are at most, and the proportion of which in Taiwan is 98%. One third of the group suffers from sleep disorder. The prevalence rate is 33.7-52%, similar with the abroad prevalence rate (38.4%), but it's much higher than the prevalence rate of the general public(20.8%). As a result, people with diabetes mellitus are at high risk of sleep disorder. Not having enough sleep or sleep badly tend to cause abnormal metabolism, which influence the control of glycemia and worsen the disease. Currently investigations emphasize prevalence rate, risk factors and diabetes mellitus, increasing glycemia, complications which result from lack of sleep. Primary improving methods include the improvement of sleeping environment, recommendation of healthy diet, exercise and getting oriental medicine treatment. At the present time, WHO is actively promoting the combination of oriental treatment. Consequently, expecting the intervention of Dao-in(Chinese Yoga) could help to improve sleep quality, HbA1c rate and oriental medicine constitution, in order to decrease the incidence of complications and improve the quality of life, which could also decrease the expense of medication and act as a health care for diabetes mellitus patients.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), diabetes is a rapidly growing chronic disease. Type II diabetes mellitus (DM) accounted for 98% of diabetics in Taiwan, and 40.0% of them have sleep disturbance similar as other country's 38.4%, but it is much higher than the people who did not have diabetics (20.8%). The metabolism and physiological status of DM patient are easily affected by poor quality of sleep, resulting in poor blood sugar control and easy to lead complications. It is a very huge impact on health. So the insomnia in DM patient is a very important care issue for medical health team. Previous studies have found that long-term practice tai chi, Ba Duan Jin and other traditional Chinese medicine qigong can improve sleep quality, glycosylated hemoglobin and physiological indicators of type 2 DM insomnia. Therefore, the aim of this study is to investigate the effect of the Duo-in on improving sleeping quality, glycated hemoglobin (HbA1c) and Traditional Chinese Medical (TCM) body constitution in insomnia of type 2 DM patient. It is expected that the results of this study could provide medical health team with reference and guidance of clinical care and home care of the patients with type 2 DM insomnia, and prevent the occurrence of complications and improve their quality of life, thereby, to reducing the cost of medical expenses.

An experimental study is designed, there will recruit 60 type 2 DM participants come from an outpatient department of a medical central in central of Taiwan, randomly assigned to experimental or control group each of 30 participants. The participants are enrolled should meet: (1) type 2 DM with diagnosis of insomnia; (2) Pittsburgh Sleep Quality Inventory Assessment score (PSQI)> 5; (3) willing to participate in and complete the consent form. The intervention method: Teach Duo-in practice (give guidance Duo-in CD disc) and the DM health education for 20 minutes in experimental group, while the control group only give the DM health education in the first 12weeks, after that the control group will give them the same intervention as experimental group for 12weeks. The experimental group performed Duo-in three times a week, each time for 20 minutes for 12 weeks at home. Daily bedtime diaries will be recorded in both groups. The tools in this study are: the scale of participant's demographic data and interference factors of sleep, PSQI, TCM body constitution questionnaire (BCQ), HbA1C and daily bedtime diaries. Data collection will be before intervention and 4th, 8th, 12th, 16th, 20th and 24th weeks, with PSQI, TCM body constitution, Glycated Hemoglobin (HbA1C) and daily bedtime diaries. The data collection on 4th, 8th, 16th and 20th week will mail the PSQI to the participants and ask them to answer. Data will analyze by descriptive and inferential statistical analysis, including frequency distribution, percentage, mean, standard deviation, Paired t-test, t-test, Chi -square test, the generalized estimation equation (GEE; to analyze the repeated measurement of different time and group) verification.

ELIGIBILITY:
Inclusion Criteria:

1. type 2 DM with diagnosis of insomnia;
2. Pittsburgh Sleep Quality Inventory Assessment score (PSQI)> 5;
3. willing to participate in and complete the consent form.

Exclusion Criteria:

* CKD
* COPD
* Mental illness
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
PSQI | 12 weeks
  Pittsburgh Sleep Quality Inventory Assessment score

SECONDARY OUTCOMES:
BCQ | 12 weeks
  body constitution questionnaire
BDNF | 12 weeks
  serum brain-derived neurotrophic factor
ABI | 12 weeks
  ankle-brachial index

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided